CLINICAL TRIAL: NCT07107685
Title: Osteoarticular Sepsis In Intensive Care Units : a Retrospective Study About Deceased Patients.
Brief Title: Prosthetic Joint Infection : Lessons From Deceased Patients in Critical Care.
Acronym: OASIS²
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250872
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Osteoarticular Infections; Intensive Care Patients; Prosthetic Joint Infection
Keywords: Osteoarticular sepsis; sepsis; osteoarticular prothetis; intensive care; critical care; prosthetic joint infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Global cohort — All deceased patients admitted to intensive care during the study period and satisfying the eligibility criteria.

SUMMARY:
This is an observational, retrospective, multicenter study based on the use of demographic, clinical and biological data from deceased patients admitted between 2018 and 2022 to critical care with a principal or associated diagnosis of joint prosthesis infection.

Data from this study will be combined with that from the OASIS study (APHP241174/ ID-RCB: 2024-A01769-38) concerning osteoarticular sepsis on prosthetic material in critical care of living patients.

The aim of this study is to improve our knowledge of the profile, care trajectories and outcomes of patients hospitalized in critical care in the context of osteoarticular material sepsis.

The results of the study could help identify at-risk populations and improve management strategies for patients with osteoarticular sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older.
* Hospitalization in critical care (intensive care unit or continuing care unit) between 2018 and 2022, lasting at least 48 hours, with a prosthetic joint infection (hip, knee, or shoulder prosthesis infection) as the primary or associated diagnosis.
* Deceased patient who had not refused data processing.

Exclusion Criteria:

* Infection involving osteosynthesis material
* Infection involving spinal instrumentation
* Patient with multiple infected prostheses
* Recurrence of prosthetic infection with the same microorganism as a previous episode
* Patient under legal protection
* Pregnant or breastfeeding patient
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients (intensive care and continuing care), admitted between 2018 and 2022 with a principal or associated diagnosis of joint prosthesis infection, who have since died.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Epidemiological description of deceased patients | 2 years
  Demographic data, medical history, history of Periprosthetic Joint Infection (timing, diagnosis, surgery, antibiotics), data in intensive care unit (leng of stay, organ failure, drugs and mechanical support, biological data) and outcome (time of death within 2 years after admission to Intensive Care Units).

SECONDARY OUTCOMES:
Composite endpoint reflecting poor clinical outcome | 2 years
  * Mortality, measured in critical care, at 30 days, 1 year and 2 years.
  * Therapeutic failure at 2 years, defined as mechanical or septic failure.
  * Functional failure at 2 years, defined as failure to resume walking and usual activities, to return home, or to regain autonomy.
Mortality at 2 years | 2 years
Epidemiological description based on the number (n) and proportion (%) of bacterial strains found in samples collected during the operation. | 2 years
  Special focus on: Gram-positive bacteria (Staphylococcus, Streptococcus, Enterococcus), Gram-negative bacteria (Enterobacteriacea, Pseudmononas), slow-growing bacteria (Cutibacterium, Corynenbacteria), yeasts; resistance mechanisms (meticillin, rifampicin, quinolone, glycopeptide, ESBL, carbapenem).

CONTACTS AND LOCATIONS:
Overall Officials: Carine PARE, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Paris, France, France

IPD SHARING:
Plan to Share IPD: No